CLINICAL TRIAL: NCT05268042
Title: Moderately Carbohydrate-restricted Diet as Treatment Targeting Improvement in Hepatic Lipid and Insulin Sensitivity in Adolescents With NAFLD
Brief Title: Moderately Carbohydrate-restricted Diet to Treat NAFLD in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Amy Miskimon Goss, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pediatric NAFLD study; R01DK128457 (NIH)
Record Dates: First submitted 2022-02-15; First posted 2022-03-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Obesity
Keywords: NAFLD; Obesity; Insulin sensitivity
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Insulin Resistance | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Intervention Model Description: The objective of this parallel arm, randomized clinical trial is to use a 6-month family-based intervention with 2 phases, a 12-week controlled feeding and 12-week free-living phase, to examine the effects of weight maintaining, moderately carbohydrate-restricted vs fat-restricted diets in adolescents with NAFLD on depletion of hepatic lipid, improvement in hepatic insulin sensitivity, and changes in the plasma metabolome.
Who Masked: Investigator, Outcomes Assessor
Masking Description: This is a dietary intervention. As such, participants will likely know what diet prescription they are randomized to during the intervention. All investigators and individuals responsible for data analysis will be blinded to participant group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Moderately carbohydrate-restricted diet (Experimental): For this study, the investigators will use the low glycemic, moderately carbohydrate-restricted diet that the investigators have previously shown is associated with depletion of hepatic lipid content, and improvement in insulin resistance in adolescents with NAFLD. This diet has a macronutrient composition of approximately 25% energy from carbohydrate, 20% energy from protein, and 55% energy from fat. No food group is excluded in this diet prescription; however, the diet emphasizes low-glycemic sources of carbohydrate, and includes mainly whole foods (vegetables, fruits, whole grains) with minimal highly processed grain products and added sugar. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements if necessary. Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included.
  Interventions: Other: Moderately carbohydrate-restricted diet
- Fat-restricted diet (Active Comparator): The fat-restricted, control diet will consist of approximately 60% carbohydrate, 20% protein, 20% fat. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables. The meal plans will minimize cholesterol, high-fat foods, high-cholesterol foods, processed starches, and added sugar, and will provide <2300 mg/day sodium. Saturated fat will be limited to 10% of total fat intake, and all dairy products will be fat-free (or low fat).
  Interventions: Other: Fat-restricted diet

INTERVENTIONS:
Other: Moderately carbohydrate-restricted diet — For this study, the investigators will use the low glycemic, moderately carbohydrate-restricted diet that the investigators have previously shown is associated with depletion of hepatic lipid content, and improvement in insulin resistance in adolescents with NAFLD. This diet has a macronutrient composition of approximately 25% energy from carbohydrate, 20% energy from protein, and 55% energy from fat. No food group is excluded in this diet prescription; however, the diet emphasizes low-glycemic sources of carbohydrate, and includes mainly whole foods (vegetables, fruits, whole grains) with minimal highly processed grain products and added sugar. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements if necessary. Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included.
  Arms: Moderately carbohydrate-restricted diet
Other: Fat-restricted diet — The fat-restricted, control diet will consist of approximately 60% carbohydrate, 20% protein, 20% fat. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables. The meal plans will minimize cholesterol, high-fat foods, high-cholesterol foods, processed starches, and added sugar, and will provide <2300 mg/day sodium. Saturated fat will be limited to 10% of total fat intake, and all dairy products will be fat-free (or low fat).
  Arms: Fat-restricted diet

SUMMARY:
This will be a 6-month randomized clinical trial with two arms: moderately carbohydrate-restricted diet and a fat-restricted control diet. This 6-month study will have 2 phases: a 12-week controlled feeding phase and a 12-week "free living" phase. During the controlled feeding phase, all food will be provided to the families of the participants for the entirety of the 12 weeks. Participants (n=80) will have been diagnosed with NAFLD based on the presence of current evidence of active disease, which will be determined by the ongoing presence of hepatic steatosis estimated by diffusely echogenic liver via ultrasound suggestive of fatty liver and a serum alanine aminotransferase (ALT) level of 45 U/L or greater. All participants will be children and adolescents age 10-17 yrs.; will have an HbA1c <7.0; and will be overweight or obese (BMI >85th percentile). It is anticipated that most participants will be sedentary. The investigators will inquire as to routine physical activity at screening. All participants will be asked to maintain their usual level of physical activity throughout the study. Physical activity will be monitored via a smart watch provided to each participant at the beginning of the study, and participants will be queried weekly by the study dietitian regarding changes in physical activity. Participants who use oral contraceptives will be asked to maintain consistent use of these preparations throughout the study. Hormone use will be examined as a potential covariate in statistical analyses.

DETAILED DESCRIPTION:
Under energy balance conditions when carbohydrates are restricted, protein or fat will increase. Large increases in dietary protein are undesirable due to the potential stimulation of hepatic gluconeogenesis. If dietary fat is increased, attention should be paid to the quality or composition of this fat. In order to minimize differences in the quality and composition of fats included in both diets, consumption of similar proportions and sources of saturated, mono-and polyunsaturated fats will be emphasized. Increased intake of polyunsaturated fats (ω-3 and ω-6) have been shown to decrease hepatic inflammation, improve hepatic function, and inhibit de novo lipogenesis; thus, diets will provide a 4:1 ratio of poly- to monounsaturated fatty acids. Because the carbohydrate-restricted diet will limit total grams of carbohydrate, total fat will increase thereby increasing the amount of dietary cholesterol provided by the diet, which may be unavoidable. However, the diet prescriptions will be matched for and provide adequate sodium intake.

carbohydrate-restricted diet. For this study, the investigators will use the low glycemic, carbohydrate-restricted diet that the investigators have previously shown is associated with depletion of hepatic lipid content, and improvement in insulin resistance in adolescents with NAFLD. This diet has a macronutrient composition of approximately 25% energy from carbohydrate, 20% energy from protein, and 55% energy from fat. No food group is excluded in this diet prescription; however, the diet emphasizes low-glycemic sources of carbohydrate, and includes mainly whole foods (vegetables, fruits, whole grains) with minimal highly processed grain products and added sugar. The investigators have successfully incorporated a limited number of "convenience" foods in our carbohydrate-restricted diet.. Incorporation of these foods increases the ultimate translatability of the carbohydrate-restricted diet, and the likelihood that participants can and will continue with the diet on their own initiative. Thus, the investigators will include some convenience foods in this study, as appropriate for the individual participant's needs. Protein foods will include meat, poultry, fish, eggs, and whey protein supplements if necessary. Fat-containing foods will include olive, coconut, and nut oils; butter; tree nuts and nut butters; cheese; cream; coconut milk; avocados; and the fat found in meat. A number of full-fat dairy products will be included. These products provide specific fatty acids that will be used to assess adherence. Saturated fat will be limited to less than 10% of daily total fat intake. Patients will obtain the majority of their fat intake from poly- and mono-unsaturated fatty acids at a 4:1 ratio (from nuts, nut butters, and from fresh fish), and saturated fat will be primarily derived from medium-chain triglycerides (e.g., coconut oil and cream), some meat, and dairy.

Fat-restricted diet. The fat-restricted, control diet will consist of approximately 60% carbohydrate, 20% protein, 20% fat. Participants will be given low-fat foods, whole-grain foods, fruits, and vegetables. The meal plans will minimize cholesterol, high-fat foods, high-cholesterol foods, processed starches, and added sugar, and will provide <2300 mg/day sodium. Saturated fat will be limited to less than 10% of total fat intake, and all dairy products will be fat-free (or low fat). Patients will obtain the majority of their fat intake from poly- and mono-unsaturated fatty acids at a 4:1 ratio matched to the carbohydrate-restricted group; however, total grams will be lower. Although the fat-restricted diet will be a high quality, healthful diet, it will include a greater amount of carbohydrate foods from such sources as bread, potatoes, and pasta that will distinguish it qualitatively from the carbohydrate-restricted diet. In addition, it will have a higher glycemic load than the carbohydrate-restricted diet. Thus, the greater glycemic load of the fat-restricted diet will derive from both inclusion of foods with a higher glycemic index and incorporation of a greater proportion of total energy from carbohydrates.

Controlled feeding phase (Phase 1) During the first 12-weeks, all food will be provided to participants. Participants will receive their weekly groceries via home delivery from a grocery store via a grocery delivery service. The study dietitian will order all groceries on-line, and the groceries will be delivered to the participants at their selected time and date. In cases where the participant's family lives outside of delivery zones, the food will be delivered to University of Alabama at Birmingham (UAB) (the Department of Nutrition Sciences' Webb Building), and the family will pick up the food during their weekly meeting with the study dietitian. This method is popular with participants, logistically feasible, and has worked very well to encourage diet adherence and attendance of study visits. Our staff has developed recipes, meal plans, and food lists that will govern the grocery selection, and will assist with implementation of the diets by providing specific meal plans and recipes. The meal plans will be prepared using Nutrition Data System for Research (NDSR), which provides a comprehensive output of diet composition including macro- and micro-nutrients, glycemic index, glycemic load, and vitamins. Meal plans may be modified after the participants become familiar with their diets, allowing for participant choice of favorite foods and meals. Based on our previous intervention, the investigators do not anticipate any difficulties with adhering to the diets for 12 weeks. Both diets will be prescribed at a weight-maintaining energy level [1.46-1.62 for females or 1.54-1.86 for males (depending on age and activity level) x measured resting energy expenditure to avoid confounding by changes in body weight. Body weight will be monitored weekly, and any participant who demonstrates consistent weight gain or loss will have their prescription revised.

Although meals will be prescribed, both diet groups will be asked to verify what they ate each week. They will be given detailed weekly meal plans in the form of a checklist, and asked to verify that each food was consumed in the prescribed amount, or to write down any deviation from the prescription.

Free living phase (Phase 2) All participants in both treatment groups will be asked to continue their assigned diet during the free-living phase when groceries are not provided. The study dietitian will work with families to devise a diet prescription that will both meet their prescribed diet guidelines and is also affordable and accessible to the families.

b.Self-monitoring: Self-monitoring of diet and exercise behaviors has repeatedly been found to be a key behavior strategy for improving adherence. Children and parents in the study will be asked to self-monitor their diet using a food recording app.

ELIGIBILITY:
Inclusion Criteria:

* clinical-pathological diagnosis of NAFLD and current evidence of active disease, which will be determined by the ongoing presence of hepatic steatosis estimated by diffusely echogenic liver via ultrasound suggestive of fatty liver and a serum alanine aminotransferase (ALT) level of 45 U/L or greater.
* age 10 -17 yrs
* overweight or obese (BMI >75th percentile).

Exclusion Criteria:

* pregnancy
* HbA1c >7%
* history of parenteral nutrition
* hepatic virus infections (HCV RNA-polymerase chain reaction negative; hepatitis A, B, C, D, E, and G; cytomegalovirus; and Epstein-Barr virus)
* use of medications known to induce steatosis (e.g. valproate, amiodarone, or prednisone), elevate liver enzymes, or affect body weight and carbohydrate metabolism (within the last 6months)
* autoimmune liver disease
* metabolic liver disease
* Wilson's disease
* genetic conditions (e.g. glycogen storage disorder) leading to hepatic steatosis;
* history of bariatric surgery
* participants and parents/guardians unwilling or unable to give informed consent, accept random assignment, attend dietary counseling sessions, adhere to treatment prescription, or complete study measures
* inability to speak and comprehend English (participants and parents/guardians)
* currently receiving intense lifestyle modification treatment
* estimated Glomerular Filtration Rate (eGFR) <60
* alcohol, tobacco or recreational drug use
* unable to undergo MRI.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Hepatic lipid | Baseline
  Hepatic lipid will be measured using MRI and Magnetic resonance spectroscopy (MRS).
Hepatic lipid | 3 months
  Hepatic lipid will be measured using MRI and MRS.
Hepatic lipid | 6 months
  Hepatic lipid will be measured using MRI and MRS.

SECONDARY OUTCOMES:
Hepatic insulin sensitivity | Baseline
  Insulin sensitivity will be measured using a euglycemic, hyperinsulinemic clamp with deuterium-labeled glucose tracers
Hepatic insulin sensitivity | 3 months
  Insulin sensitivity will be measured using a euglycemic, hyperinsulinemic clamp with deuterium-labeled glucose tracers
Plasma metabolome | Baseline
  Metabolomic profile will be assessed from a fasted blood sample.
Plasma metabolome | 3 months
  Metabolomic profile will be assessed from a fasted blood sample.
Body composition | Baseline
  Body composition will be assessed using Dual energy X-ray absorptiometry
Body composition | 3 months
  Body composition will be assessed using Dual energy X-ray absorptiometry
Body composition | 6 months
  Body composition will be assessed using Dual energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States